CLINICAL TRIAL: NCT00497224
Title: Phase II Trial of Erlotinib in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-Tar-725
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Cancer; Pancreas
Keywords: Pancreatic Cancer; Pancreatic Carcinoma; Pancreas; Adenocarcinoma; Erlotinib; Tarceva; OSI-774; Phase II
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Adenocarcinoma | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental): Eligible patients will receive erlotinib 150mg PO daily, with dose escalation occurring as tolerated.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib starting at 150 mg PO (by mouth) daily. Dose may increase or decrease by the study doctor as per protocol (study plan).
  Other Names: TARCEVA; OSI-774

SUMMARY:
This is an open-label, multi-center phase II study of erlotinib in patients with metastatic or locally advanced, unresectable pancreatic cancer who have received up to one line of gemcitabine based chemotherapy.

DETAILED DESCRIPTION:
Erlotinib in addition to gemcitabine significantly improves overall survival compared to gemcitabine alone in advanced pancreatic cancer (median overall survival 6.24 vs 5.91 months respectively). However, combined therapy has not become standard of care due to the modest absolute benefit. In NSCLC, the optimal efficacy of erlotinib is not in combination with first-line cytotoxic chemotherapy for advanced disease, but as a single agent after cytoxic chemotherapy. Preclinical and clinical data suggest that erlotinib will have activity as a single agent in advanced pancreatic cancer. The presence of an erlotinib-induced rash is associated with improved survival in phase II and III trials of diverse tumor types (reviewed by Perez-Soler et al.), and is associated with higher steady state concentrations of erlotinib.

This phase II trial aims to determine the safety and efficacy of erlotinib in patients with advanced pancreatic cancer who have previously been treated with up to one prior line of gemcitabine based chemotherapy for advanced disease. In addition, we will evaluate the feasibility and activity of dose escalation of erlotinib in patients who do not develop a rash. Clinical outcome will be correlated to EGFR status based on immunohistochemistry and gene amplification status as well as Kras mutations from archival tumor tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed pancreatic carcinoma that is locally advanced, unresectable or metastatic.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
* Previous therapy:

Surgery: Previous surgery is permissible. Patients must be > 4 weeks from any major surgery.

* Chemotherapy: Patients may have received up to 1 prior line of gemcitabine based systemic therapy (single agent or combination therapy) for locally advanced or metastatic disease. Prior therapy with inhibitors of angiogenesis is permitted. All toxicities must be resolved to < Grade 1 (CTCAE v 3.0) and the last dose must have been given at least 4 weeks prior to randomization.
* Patients may also have received prior 5 FU (+/- folinic acid) or gemcitabine given concurrently with radiation as a "radiation sensitizer". All toxicities must be resolved and the last dose of chemotherapy must have been given at least 4 weeks prior to randomization.
* Radiation: Patients may have received prior radiation treatment for management of local disease providing that disease progression has been documented (either locally or systemically), all toxicities have resolved, and the last fraction of radiation treatment was completed at least 4 weeks prior to randomization.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of erlotinib in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
* Life expectancy of greater than or equal to 3 months.

ECOG performance status <2.

* Patients must have normal organ and marrow function as defined below:

  * Leukocytes >/= 3,000/mcL
  * Absolute neutrophil count >/= 1,000/mcL
  * Platelets >/= 100,000/mcL
  * Total bilirubin </= 1.5 UNL
  * AST(SGOT) </= 2.5 X institutional upper limit of normal
  * INR </= 1.5 unless on warfarin (see 3.1.9)
  * Creatinine within normal institutional limits OR
  * Creatinine clearance >/= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Since CYP3A4 appears to be the major enzyme responsible for the human hepatic metabolism of erlotinib in vitro, the concurrent use of inhibitors and inducers of CYP3A4 are prohibited during the study treatment period. Concurrent use of CYP3A4 substrates are allowed, however, use caution and monitor the patient for potential drug interactions.
* There is a potential interaction between erlotinib and warfarin. Patients have experienced elevated INRs and bleeding with this combination of drugs. Patients on warfarin with PT INR >1.5 are eligible provided that all of the following criteria are met:
* The patient is therapeutic on a stable dose of warfarin
* The upper target for INR is no greater than 3.
* The patient has no active bleeding or pathological condition that carries a high risk of bleeding (e.g., CT evidence of tumor invading the duodenum or known varices).

Note: anticoagulation with low molecular weight heparin is permitted.

* The effects of erlotinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients receiving any other investigational agents concurrently are ineligible.
* Prior therapy with inhibitors of the EGFR (eg. cetuximab, EMD 72000, panitumumab, gefitinib, erlotinib) or multitargeted agents that inhibit EGFR (eg. ZD6474, AEE788).
* Patients with allergies to or a history of allergic reactions attributed to any other compound of similar chemical or biologic composition to erlotinib.
* Patients with greater than grade 1 diarrhea at baseline. Patients with pancreatic cancer often have diarrhea due to pancreatic insufficiency, so a trial of pancreatic enzymes may be warranted to reduce baseline diarrhea.
* PT INR >1.5 unless the patient is on full-dose warfarin.
* Patients with any condition that impairs their ability to swallow and retain pills
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because erlotinib has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with erlotinib, breastfeeding should be discontinued if the mother is treated with erlotinib.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with erlotinib. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-11; Primary Completion 2008-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | Clinically assessed every cycle (month) and radiologically assessed every 2 cycles (2 months) with CT scan
  Measured by the rate of disease control (objective response plus prolonged stable disease), in patients with unresectable, locally advanced or metastatic pancreatic adenocarcinoma.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability of Erlotinib] | Assessed every cycle (month)
  Incidence of adverse events related to treatment, through monthly SAE analysis.
Tolerability of Erlotinib Dose Escalation | assessed cycle 1, day 28, then every cycle (month)
  Assessment erlotinib dose escalation efficacy through analysis of patients who do not develop a rash by cycle 1, day 15.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Moore, MD, Principal Investigator — Drug Development Program, Princess Margaret Hospital
Locations (5):
- Canada (5):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Renouf DJ, Tang PA, Hedley D, Chen E, Kamel-Reid S, Tsao MS, Tran-Thanh D, Gill S, Dhani N, Au HJ, Wang L, Moore MJ. A phase II study of erlotinib in gemcitabine refractory advanced pancreatic cancer. Eur J Cancer. 2014 Jul;50(11):1909-15. doi: 10.1016/j.ejca.2014.04.008. Epub 2014 May 21. PMID 24857345